CLINICAL TRIAL: NCT06404255
Title: Evaluating the Impact of a Stress Management Training Course for ECOS Preparation for Medical Students
Brief Title: Impact of a Stress Management Training Course
Acronym: FORSE
Status: Not yet recruiting | Type: Observational
Sponsor: Université Paris-Saclay (Other)
Responsible Party: Principal Investigator, Guillemette Fouquet, Prinicipal investigator, Université Paris-Saclay
Other Study IDs: FORSE_001
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical students: Medical students from the University of Paris-Saclay, during hospital internships Stress assessement with or without a stress management training
  Interventions: Behavioral: Stress management training

INTERVENTIONS:
Behavioral: Stress management training — Stress management training

SUMMARY:
Objective structured clinical examinations (ECOS) are playing an increasingly important role in the training and assessment of medical students, and now account for 30% of the grade for access to the 3rd cycle of medical studies.

Although students generally seem to have a favorable opinion of this examination modality, several studies have reported that ECOS are a greater source of stress than other types of examination, particularly written examinations.

The investigators aim to assess the benefits of a stress management training for medical students, on the negative impact of stress during ECOS.

The investigators hypothesize that training in stress management could be beneficial for medical students, in particular to prepare them mentally to limit the negative impact of stress durgin ECOS, and ultimately reduce their overall stress and potentially improve their performance.

DETAILED DESCRIPTION:
Objective structured clinical examinations (ECOS) are playing an increasingly important role in the training and assessment of medical students, and now account for 30% of the grade for access to the 3rd cycle of medical studies.

Although students generally seem to have a favorable opinion of this examination modality, several studies have reported that ECOS are a greater source of stress than other types of examination, particularly written examinations.

Anxiety can affect students' performance, although not all studies have found a significant correlation between results and students' state of anxiety.

However, it is essential to take account of students' well-being, especially as it has been shown that medical students suffer from symptoms of anxiety and depression, some of which may be related to their studies.

It is therefore important to reduce these symptoms of anxiety in order to improve students' well-being, and eventually their performance during ECOS.

A number of studies have looked at ways of reducing student anxiety, including breathing relaxation techniques and anxiety management programs. Preparation, stress management and self-confidence can have a calming effect, and may even have a positive impact on exam performance.

The visual analog stress scale and the STAI questionnaire are two validated and commonly used methods for stress assessment. The investigators modified the visual scale to assess the functional impact of stress on ECOS performance.

The investigators hypothesize that training in stress management could be beneficial for medical students, in particular to prepare them mentally to limit the negative impact of stress durgin ECOS, and ultimately reduce their overall stress and potentially improve their performance.

The investigators aim to assess the benefits of a stress management training for medical students, on the negative impact of stress during ECOS.

ELIGIBILITY:
Inclusion Criteria:

* Medical students from Paris Saclay University, during hospital internships
* Agreeing to take part in the study

Exclusion Criteria:

* Refusal to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical students from Paris Saclay University, during hospital internships
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Functional impact of stress after ECOS | 3 years
  Score for the functional impact of stress after ECOS, with or without stress management training From 0 = No negative impact of stress on ECOS performance To 10 = Extremely negative impact of stress on ECOS performance

SECONDARY OUTCOMES:
Anxiety score | 3 years
  Anxiety score on STAI (State and Trait Anxiety Inventory) after ECOS, with or without stress management training From 0 = no anxiety To 40 = very high anxiety
ECOS scores | 3 years
  ECOS scores, with or without stress management training From 0 = lowest score To 10 = highest score

IPD SHARING:
Plan to Share IPD: Undecided